CLINICAL TRIAL: NCT06373497
Title: IT2023-08-ATKINS-ATHERO-RT: Real-Time Atherosclerosis Activity After Thoracic Radiotherapy Using Sodium Fluoride Positron Emission Tomography
Brief Title: Real-Time Atherosclerosis Activity After Thoracic Radiotherapy Using Sodium Fluoride Positron Emission Tomography
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Katelyn Atkins (Other)
Responsible Party: Sponsor-Investigator, Katelyn Atkins, Sponsor-Investigator, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023-08-ATKINS-ATHERO-RT
Record Dates: First submitted 2024-04-11; First posted 2024-04-18 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Oligometastatic Disease
Keywords: Thoracic Radiotherapy; PET Imaging; MRI Imaging; 18 F-NaF; Clinical Stage II; Clinical Stage III

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Fluorine-18-sodium fluoride (18F-NaF) PET/MRI imaging with CT angiography
  Interventions: Diagnostic Test: 18-F-NaF Cardiac PET/MRI and; Diagnostic Test: CT Angiogram

INTERVENTIONS:
Diagnostic Test: 18-F-NaF Cardiac PET/MRI and — All eligible subjects will receive 18-F-NaF Cardiac PET/MRI at baseline and 6 months after the completion of radiotherapy where the heart is in the treatment field
Diagnostic Test: CT Angiogram — All eligible subjects will receive CT Angiogram at baselin

SUMMARY:
The prospective single-arm pilot study, ATHERO-RT: Real-Time Atherosclerosis Activity after Thoracic Radiotherapy using Sodium Fluoride Positron Emission Tomography, will aim to:

1. To deploy first-in-kind application of fluorine 18-sodium fluoride (18F-NaF) PET (Positron Emission Tomography) /MRI (Magnetic Resonance Imaging) imaging to detect real-time atherosclerosis activity at the time of cancer diagnosis and after cardiac radiation exposure
2. To detect longitudinal changes in clonal hematopoiesis (CH) genetic architecture following thoracic RT (Radiation Therapy) in patients at high risk of cardiac dysfunction, and
3. To measure perturbations in the immune-modulatory and metabolic states following thoracic RT (Radiation Therapy) exposure in patients at high risk of cardiac dysfunction.

Eligible patients will be adults (≥18 years old) with Stage II-III or oligo-metastatic stage IV malignancy (any histology) at high risk for RT-associated cardiac toxicity (defined as receiving ≥30 Gy (Gray) RT where the heart is in the treatment field54). The study will enroll a total of 10 subjects, recruited from Cedars-Sinai Medical Center. The primary endpoint will be successful completion of 18F-NaF PET imaging at the baseline and 6-month post-RT time points. Blood will be collected at baseline, end of RT, and 6-months post-RT.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years.
* Have clinical stage II-III or oligo-metastatic stage IV malignancy (any histology) planned to be treated with thoracic radiotherapy (≥30 Gy) where the heart is in the treatment field.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2.
* Planning to receive standard of care radiotherapy treatment.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
* Ability to read, write, and understand English

Exclusion Criteria

* Estimated glomerular filtration rate (eGFR) <45 mL/min/m2 or serum creatinine ≥1.5 mg/dL.
* Patients with a known or previous allergy to iodinated contrast, gadolinium contrast, and/or 18F-NaF tracer.
* Inability to receive PET tracer.
* Inability to receive MRI, requiring sedation for MRI, or prohibitive implant and/or device, including ferromagnetic implants and ferromagnetic foreign bodies.
* Subjects with claustrophobia, problems being in enclosed spaces, or inability to lie supine.
* Subjects that are pregnant or breastfeeding.
* Subjects unable to comply with visit instructions, including inability to lie still, hold breathe, or follow procedure instructions.
* Allergy to animal dander or animal-instigated asthma.
* Any other condition which, in the opinion of the investigator, may make the patient a poor candidate for participation in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using F-NaF PET/MRI imaging | 6 Months
  To determine the feasibility of using 18F-NaF PET/MRI imaging for detection of real-time atherosclerosis activity in patients at high risk of RT-associated cardiac dysfunction.

SECONDARY OUTCOMES:
Incidence of MACE | One Year
  To measure the one-year cumulative incidence of MACE (Major Adverse Cardiovascular Events). The one-year cumulative incidence of MACE will be estimated, adjusting for non cardiac death as a competing risk. For the secondary endpoint, one-year MACE cumulative incidence will be estimated using the Cumulative Incidence Function (CIF), while accounting for non-cardiac death as a competing risk.

CONTACTS AND LOCATIONS:
Overall Officials: Katelyn Atkins, MD, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No